CLINICAL TRIAL: NCT01398397
Title: Medical Record Review of Hypohidrotic Ectodermal Dysplasia Clinical Phenotype
Acronym: ECP-006
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Collaborators: National Foundation of Ectodermal Dysplasia (Unknown)
Responsible Party: Sponsor
Other Study IDs: ECP-006
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Hypohidrotic Ectodermal Dysplasia; X-Linked Hypohidrotic Ectodermal Dysplasia
Keywords: HED; XLHED; X-linked Hypohidrotic Ectodermal Dysplasia (XLHED)
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to collect information about people who have or may have Hypohidrotic Ectodermal Dysplasia (HED) or X-linked Hypohidrotic Ectodermal Dysplasia (XLHED). This study will allow Edimer Pharmaceuticals to know more about HED/XLHED so that hopefully the investigators can develop a drug to treat this condition. In this study Edimer will retrospectively review and abstract (summarize) medical records of people that have or may have HED/XLHED in order to further understand the natural history and disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

-Males or females with:

1. the clinical characteristics of HED, including at least two of the following characteristics: a history of decreased sweating;abnormal teeth (fewer permanent teeth, teeth are smaller than average and often have conical crowns);sparseness of scalp and body hair.

   -OR-
2. genetically confirmed HED or XLHED;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll up to fifty HED/XLHED affected individuals.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-04

CONTACTS AND LOCATIONS:
Locations (1):
- Edimer Pharmaceuticals, Cambridge, Massachusetts, United States